CLINICAL TRIAL: NCT00858533
Title: A Pilot Controlled Feasibility Trial of Early Health At Work Workplace Intervention
Brief Title: Trial of Health At Work Workplace Health Intervention
Acronym: H@W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BER10457
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2010-01

CONDITIONS: Workplace Health
Keywords: early intervention; sickness absence; return to work; primary care
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- workplace health advice (Other): The intervention group will receive additional support from a H@W Workplace Health Advisor who will deliver an intervention aimed at sickness absence prevention or sustained return to work, depending on individual circumstances.
  Interventions: Behavioral: Health at Work workplace health advice and support
- GP sickness absence consultation (No Intervention): Routine general practitioner care for workplace sickness absence.

INTERVENTIONS:
Behavioral: Health at Work workplace health advice and support — The intervention group will receive additional support from a H@W Workplace Health Advisor who will deliver an intervention aimed at sickness absence prevention or sustained return to work, depending on individual circumstances. The intervention will be standardized as far as possible to show types of activity undertaken with participants, their GP, line managers, human resources departments and trade union representatives.
  Arms: workplace health advice

SUMMARY:
This pilot study will compare workplace health intervention delivered by advisors based in GP practices with normal GP care to assess the usefulness of the concept and its potential for wider use in a larger randomised controlled trial.

DETAILED DESCRIPTION:
The aim of this pilot study is to examine the impact of H@W intervention(s) on job retention and return to work and compare outcomes with those from normal GP care. The target population for this study is people still at work but experiencing a work-related health problem as well as those off work. For the purpose of the study, short term sickness absence is defined as a period of 4 weeks or less and long term sickness absence defined as a period of 4 weeks or longer. Hypothesis

That H@W intervention in comparison to standard care:

* promotes work retention
* enables a quick and sustained return to work for those on short term sick leave (4 weeks or less)
* achieves sustained return to work for those on long term sick leave of 4 weeks or more. This could include a phased return to work.
* achieves positive outcomes which could mean leaving one job and starting another.

ELIGIBILITY:
Inclusion Criteria:

* People with work related health problems registered with GP practices in Liverpool Primary Care Trust.

Exclusion Criteria:

* People registered with GP practices outside Liverpool Primary Care Trust.
* Vulnerable adults and those considered by their GP to be unsuitable for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of days off work through sickness absence after index consultation, which will also apply to people at work with a work-relevant condition | 1 year

SECONDARY OUTCOMES:
Secondary outcome measure: time to first return to work (RTW) allowing for phased return. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Gabbay, MD, Principal Investigator — University of Liverpool
Locations (1):
- Division of Primary Care, University of Liverpool., Liverpool, Merseyside, United Kingdom